CLINICAL TRIAL: NCT04360343
Title: A Randomized, Open-label, Single Dose, 2-period, 2-sequence, 2-treatment, Crossover Study to Compare the Pharmacokinetics, Pharmacodynamics and Safety/Tolerability of LC51-0255 Film-coated Tablet (SG85) With LC51-0255 Uncoated Tablet (SG82) in Healthy Subjects
Brief Title: Compare the Pharmacokinetics, Pharmacodynamics and Safety/Tolerability of LC51-0255 Film-coated Tablet (SG85) With LC51-0255 Uncoated Tablet (SG82) in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: LG-SGCL003
Record Dates: First submitted 2020-04-06; First posted 2020-04-24 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- LC51-0255 film-coated tablet (Experimental): Drug: LC51-0255
  Interventions: Drug: Film-coated tablet
- LC51-0255 uncoated tablet (Active Comparator): Drug: LC51-0255
  Interventions: Drug: Film-coated tablet

INTERVENTIONS:
Drug: Film-coated tablet — uncoated tablet

SUMMARY:
To compare the pharmacokinetics, pharmacodynamics and safety/tolerability of LC51-0255 film-coated tablet (SG85) with LC51-0255 uncoated tablet (SG82) in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females between the age of 19 and 45 at the screening visit
2. Subjects with the Body Mass Index (BMI) measurement results between 18.0 kg/m2 and 27.0 kg/m2 at the screening visit
3. Subjects who were confirmed to be healthy based on the medical history
4. Subjects who make a voluntary decision to participate in this clinical study and provide the informed consent

Exclusion Criteria:

1. Subjects with a clinically significant disease or history in liver, kidney, gastrointestinal system, respiratory system, musculoskeletal system, endocrine system, neuropsychiatric system, hemato-oncology system or cardiovascular system
2. Subjects with a disease (e.g., Crohn's disease, etc.) or history of surgery (except for simple appendectomy and herniotomy) in gastrointestinal system which may affect the absorption of the investigational product
3. Subjects with a history of clinically significant disease or suspicious sign/symptom of ophthalmologic disease including uveitis and retinitis at the screening visit
4. Subjects who had donated whole blood within 2 months, component blood within 1 month, or received transfusion within 1 month prior to the first administration day
5. Subjects who had taken an inducer or inhibitor of drug metabolism such as barbiturates etc. within 1 month prior to the first administration day
6. Subjects who had eaten grapefruit/caffeine-containing food within 3 days prior to the first hospitalization or subjects who could not stop taking food containing grapefruit or caffeine from 3 days prior to hospitalization to the discharge day
7. Subjects who had taken any prescription drug or herbal medicine within 2 weeks or any over the counter (OTC) drug within 1 week prior to the first administration day (however, subjects fulfilling other conditions could participate in the study at the investigator's discretion)
8. Subjects who taking excessive caffeine or alcohol or heavy smoker (caffeine > 5 units/day, alcohol > 21 units/week (1 unit = 10 mL as pure alcohol), smoking > 10 cigarettes/day)
9. Subjects who had a history of tuberculosis (TB) infection or a positive result in the Quantiferon TB-Gold test and the chest X-ray in the screening tests
10. Subjects who unable to take the food provided by the study institution
11. Subjects who with a positive result in the serology test (hepatitis B test, human immunodeficiency virus (HIV) test, hepatitis C test, syphilis test)
12. Other cases that the investigator consider unsuitable as the subject

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic Outcome Measures | baseline,during the procedure
  Peak Plasma Concentration (Cmax)
Pharmacokinetic Outcome Measures | baseline,during the procedure
  Area under the plasma concentration versus time curve (AUC)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University College of Medicine and Hospital, Seoul, South Korea